CLINICAL TRIAL: NCT02889601
Title: Psycho-behavioral Disorders in Frontotemporal Lobar Degeneration: Validation of a Quantification and Follow-up Scale
Brief Title: DAPHNE Scale Validation in Frontotemporal Lobar Degeneration
Acronym: DAPHNE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_0463
Record Dates: First submitted 2016-08-24; First posted 2016-09-05 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Frontotemporal Lobar Degeneration
MeSH Terms: conditions — Frontotemporal Lobar Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fronto-temporal lobar degeneration: DAPHNE score building and internal validation through Fronto-temporal lobar degeneration patients.
  Interventions: Other: Psycho-behavioural assessment
- Control: External validation of DAPHNE score among patients with Alzheimer's disease, progressive supranuclear palsy and bipolar disorder with cognitive disorders.
  Interventions: Other: Psycho-behavioural assessment

INTERVENTIONS:
Other: Psycho-behavioural assessment — DAPHNE Scale

SUMMARY:
Psycho-behavioral disorders assessment is crucial for the diagnosis and follow-up of patients with frontotemporal degeneration (FTD). DAPHNE scientific staff have therefore developed a quantification and follow-up scale specifically dedicated to patients with FTD in current clinical practice. This scale is called DAPHNE to Disinhibition, Apathy, Perseveration, Hyper orality, Negligence and loss of Empathy.

DETAILED DESCRIPTION:
Psycho-behavioral disorders assessment is crucial for the diagnosis and follow-up of patients with frontotemporal degeneration (FTD). DAPHNE scientific staff have therefore developed a quantification and follow-up scale specifically dedicated to patients with FTD in current clinical practice. This scale is called DAPHNE to Disinhibition, Apathy, Perseveration, Hyperorality, Negligence and loss of Empathy. This study aims to validate this scale. This validation will include methodological steps required to develop a new clinical tool, by studying internal consistency, loyalty, and concurrent validity in comparison with validated existing tools. Complementarily, sensitivity and specificity will be assessed via a control population including patients with Alzheimer's disease, , progressive supranuclear palsy and bipolar disorder with cognitive disorders.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

1. Patients with FTD according Neary (1998) and Raskowsky (2011) diagnostic criteria.
2. Mini-Mental State Examination ≥ 18
3. Consent

Group 2 Control:

1. Patients with Alzheimer's disease (MacKahn, 2011), patients with supranuclear palsy (Litvan, 1996) and patients with bipolar disorder with cognitive disorders.

   criteria.
2. Mini-Mental State Examination ≥ 18
3. Consent

Exclusion Criteria:

* Minor patient

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Frontotemporal lobar degeneration according Neary (1998) and Raskowsky (2011) diagnostic criteria.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Internal validation of DAPHNE Score | Baseline
  Face validity - Structural validity - Convergent Validity - Known-groups validity - Responses consistency - Reliability

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France